CLINICAL TRIAL: NCT01692002
Title: Development of Orally Administered Sodium Propionate to Treat and Prevent Diabetes
Brief Title: Oral Propionate to Treat and Prevent Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The person who was running the study never completed it, as the study never reached the target recruitment levels.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CRO2020
Record Dates: First submitted 2012-09-11; First posted 2012-09-25 (Estimated); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Propionate
MeSH Terms: conditions — Diabetes Mellitus | interventions — sodium propionate; Sodium Chloride; Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: the study was terminated so data were referred to only 6 people despite a target recruitment of 12
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium chloride pill (Placebo Comparator): Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Interventions: Dietary Supplement: Sodium Chloride; Procedure: Oral glucose tolerance test; Procedure: Intravenous glucose tolerance test.
- Sodium propionate pill (Experimental): Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Interventions: Dietary Supplement: Sodium propionate; Procedure: Oral glucose tolerance test; Procedure: Intravenous glucose tolerance test.

INTERVENTIONS:
Dietary Supplement: Sodium propionate — Sodium propionate capsule or tablet
  Arms: Sodium propionate pill
Dietary Supplement: Sodium Chloride — Placebo capsule or tablet
  Arms: Sodium chloride pill
Procedure: Oral glucose tolerance test
Procedure: Intravenous glucose tolerance test.

SUMMARY:
The aim of these studies is to firstly determine the pharmacokinetic profile of orally administered enteric coated sodium propionate. Subsequently, the most efficacious dose at improving glucose tolerance following an oral glucose challenge will be determined. The investigators will then determine the mechanism of action of propionate, whether it acts by altering beta cell function directly or by augmenting the incretin effect or both

DETAILED DESCRIPTION:
The NHS spends £1M per hour, 10% of its yearly budget, treating diabetes. In the UK cases of diabetes are expected to top 4 million by 2025. There is an urgent need for new therapies. The short chain fatty acid propionate is a natural substance produced by digestion of fermentable carbohydrates. Preclinical and early human data demonstrate it improves pancreatic function and glucose control. The investigators aim to conduct proof of principle studies to determine if oral delivery of propionate improves glucose control in patients at risk of developing diabetes.

ELIGIBILITY:
Inclusion Criteria:

Study 1: Healthy men and women aged between 18 and 70 years with BMI between 20-25 kg/m2 and with normal fasting blood glucose (below5.5mmol/l and HbA1C less than 5.7% will be eligible to volunteer.

Study 2: As for Study 1. Study 3: Cohort 1: Volunteers aged between 30 to 70 with a BMI between 25-35 kg/m2 who do not have impaired fasting glucose and have HbA1c below 5.7%.

Cohort 2: Volunteers aged between 30 to 70 years with a BMI between 25-35 kg/m2 who have impaired fasting glucose (between 5.5-7mmol/l) and HbA1C between 5.7% and 6.5%,

* Exclusion Criteria:• Type 1 or Type 2 Diabetes

  * Gained or lost ≥ 3kg weight in the past three months
  * Taken prescription medicines having an impact on metabolism, appetite regulation, glucose homeostasis and hormonal regulation
  * Taken any dietary supplements in the last 6 months
  * Any chronic illness
  * Cardiovascular disease
  * Excess alcohol intake
  * Current smokers
  * Any gastrointestinal disorder e.g. Crohn's disease, coeliac disease or irritable bowel syndrome
  * A history of drug or alcohol abuse in the last 2 years
  * Pregnancy (all women of child bearing age will undergo a pregnancy test).
  * Pancreatitis
  * Use of medications likely to interfere with glucose metabolism, appetite regulation, hormonal balance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin A Bewick, PhD., Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Hammersmith Hospital, London, UK
  - Imperial College London, London
  - St John McMichael Centre - Imperial College London, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started March 2013 and ended August 2016. The study was based at the clinical research facility at Imperial College Health Care Trust but never completed. Only 6 where recriuted and completed. The target was 12
Pre-assignment Details: Wash out of 7 days between interventions
Groups:
- Sodium Chloride Pill: Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Sodium Chloride: Placebo capsule or tablet
  Oral glucose tolerance test
  Intravenous glucose tolerance test.
- Sodium Propionate Pill: Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Sodium propionate: Sodium propionate capsule or tablet
  Oral glucose tolerance test
  Intravenous glucose tolerance test.
Period: 1st Period of the Cross-over Study
Arm/Group | Sodium Chloride Pill | Sodium Propionate Pill
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Sodium Chloride Pill | Sodium Propionate Pill
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: 2nd Period of the Cross-over Study
Arm/Group | Sodium Chloride Pill | Sodium Propionate Pill
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: only 6 where recriuted and completed
Groups:
- Sodium Chloride: Sodium Chloride Pill Intervention
- Sodium Propionate: Sodium propionate pill
- Total: Total of all reporting groups
Arm/Group | Sodium Chloride | Sodium Propionate | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 dropped out
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 dropped out
  Participants
    Female | 2 | 2 | 4
    Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 dropped out
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 3 | 3 | 6
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 3 dropped out
  Participants
    United Kingdom | 3 | 3 | 6
Propionate [Mean (Standard Deviation); unit: micromol/l] — Population: 3 dropped out
  micromol/l | 0.05 (0.05) | 0.05 (0.05) | 0.05 (0.05)

OUTCOME MEASURES:

1. Primary Outcome: Propionate CMax
Description: Study 1: Peak plasma concentration of propionate. Dose ranging and pharmacokinetic profile of propionate by Mass spectrometry has been measured at -10, 0, 15, 30, 60, 90, 120, 150, 180, 4h, 6h, 8h (the mean below was estimated first per patient (across all the above time points) and then per arm across the 6 patients)
Time Frame: hours (up to 8hrs)
Population: Propionate concertation in plasma
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Sodium Chloride Capsule: Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Sodium Chloride: Placebo capsule or tablet
  Oral glucose tolerance test
  Intravenous glucose tolerance test.
- Sodium Propionate Capsule: Study 1: pharmacokinetics Study2: Oral glucose tolerance test Study 3: intravenous glucose tolerance test
  Sodium propionate: Sodium propionate capsule or tablet
  Oral glucose tolerance test
  Intravenous glucose tolerance test.
Arm/Group | Sodium Chloride Capsule | Sodium Propionate Capsule
Number analyzed (Participants) | 3 | 3
mmol/l | 7.2 (0.26) | 7.79 (0.25)

2. Secondary Outcome: Total Amount of Insulin Stimulated by Propionate Per Unit Time (Incremental Area Under the Curve)
Description: Study 3: Participants will undergo a frequently sampled oral glucose tolerance test (OGTT) to detect changes in insulin sensitivity and beta cell function. Where maximum insulin increments during a glucose tolerance test will be reported on a scale 0 to 1000 where 0 is the lowest and 1000 is the highest outcome
Time Frame: 10 minutes
Measure: Mean (Standard Error); unit: uM/min
Arm/Group | Sodium Chloride Capsule | Sodium Propionate Capsule
Number analyzed (Participants) | 3 | 3
uM/min | 677.5 (24) | 678 (25)

3. Secondary Outcome: Insulinogenic Index (Change in Insulin Divided by the Change in Glucose Over the First 30 Minutes of the Test)
Description: Study 2: insulinogenic index. Oral glucose tolerance dose finding was measured with commercially available kits (the mean below was estimated per arm across the 6 patients)
Time Frame: 30mins
Population: This index is estimated on a scale 0 to 50 where 0 is the lowest value and 50 is the highest value
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sodium Chloride Capsule | Sodium Propionate Capsule
Number analyzed (Participants) | 3 | 3
index | 30.2 (12) | 31 (12.5)

4. Secondary Outcome: Insulin Levels in Response to the Absorption of Proprionate (Total Insulin Across All Time Points)
Description: Plasma insulin has been measured using commercially available kits at -10, 0, 15, 30, 60, 90, 120, 150, 180, 4h, 6h, 8h (the mean below was estimated first per patient (across all the above time points) and then per arm across the 6 patients)
Time Frame: hours (up to 8 hours)
Population: The mean below was estimated first per patient (across all the above time points) and then per arm across the 6 patients.
Measure: Mean (95% Confidence Interval); unit: uM/l
Arm/Group | Sodium Chloride Capsule | Sodium Propionate Capsule
Number analyzed (Participants) | 3 | 3
uM/l | 8142 [6809 to 9737] | 8316 [7148 to 9674]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Sodium Chloride Pill | Sodium Propionate Pill
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT01692002/Prot_SAP_000.pdf